CLINICAL TRIAL: NCT01842763
Title: French Database of Occipital Nerves Stimulation in the Treatment of Refractory Chronic Headache Disorders
Acronym: NGO
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 12-PP-08
Record Dates: First submitted 2013-03-22; First posted 2013-04-30 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Refractory Chronic Headache Disorders
Keywords: Chronic daily headache; treated by occipital nerves stimulation; peripheral neuromodulation; occipital nerves; network; database
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this non interventional research is to set up a French database, initially for 3 years, of patients suffering from refractory chronic headache disorders (chronic migraine, cluster headache, chronic paroxysmal hemicranias, SUNCT syndrome, hemicrania continua, cervicogenic headache disorders), and treated by occipital nerves stimulation.

Every team using this neuromodulation approach in France is likely to participate in the network.

Fifty patients a year are expected. They will be informed about data which are collected and why they are collected.

The data will come from medical files and questionnaires filling out by the patients. The data will be collected on a case report form adapted to each refractory chronic headache disorder. The case report form pages will be faxed to the coordinating team who will enter the data in the database and analyse the data in a descriptive manner.

These data are social and demographic data, medical data (headache features, headache functional and emotional impact, medications, and concomitant medical conditions), technical data (kind of electrodes and implantable pulse generator used, stimulation parameters chosen), and safety data.

This research should provide an update on practices, an evaluation of the efficacy and long term safety of occipital nerves stimulation, and perhaps help in identifying response predictive factors to this neuromodulation approach.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from refractory chronic headache disorders and treated by occipital nerves stimulation

Exclusion Criteria:

* patients who don't agree with participating in the study because the ending of professional confidentiality is required for setting up the database

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from refractory chronic headache disorders (chronic migraine, cluster headache, chronic paroxysmal hemicranias, SUNCT syndrome (Short-lasting Unilateral Neuralgiform headache attacks with Conjunctival injection and Tearing), hemicrania continua, cervicogenic headache disorders) according to ICHD-II
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
observation of a disease or medical condition under normal conditions | at each visit (up to 4 years)
  social and demographic data, medical data (headache features, headache functional and emotional impact, medications, and concomitant medical conditions), technical data (kind of electrodes and implantable pulse generator used, stimulation parameters chosen), and safety data.

CONTACTS AND LOCATIONS:
Overall Officials: Michel LANTERI-MINET, Principal Investigator — CHU de Nice département d'évaluation et traitement de la Douleur
Locations (16):
- France (16):
  - Hopitaux Civil de Colmar, Colmar, Haut-rhin
  - Clermont Ferrand CHU, Clermont-Ferrand
  - Annecy Genevois CHU, Épagny
  - Grenoble CHU, Grenoble
  - Lille CHU, Lille
  - Limoges CHU, Limoges
  - HCL, Lyon
  - APHM, Marseille
  - Nancy CHU, Nancy
  - Nantes CHU, Nantes
  - Département d'Evaluation et Traitement de la Douleur, Nice
  - AP-HP Lariboisière, Paris
  - Adolphe de Rothschild Foundation, Paris
  - Poitiers CHU, Poitiers
  - Saint Etienne CHU, Saint-Etienne
  - Foch Hospital, Suresnes

REFERENCES:
- [Derived] Balossier A, Donnet A, Regis J, Leplus A, Lanteri-Minet M, Fontaine D. Occipital Nerve Stimulation for Recurrent Trigeminal Neuralgia Without Occipital Pain. Neuromodulation. 2023 Dec;26(8):1795-1801. doi: 10.1016/j.neurom.2022.03.012. Epub 2022 Jun 7. PMID 35688701
- [Derived] Fontaine D, Blond S, Lucas C, Regis J, Donnet A, Derrey S, Guegan-Massardier E, Jarraya B, Dang-Vu B, Bourdain F, Valade D, Roos C, Creach C, Chabardes S, Giraud P, Voirin J, Bloch J, Rocca A, Colnat-Coulbois S, Caire F, Roger C, Romettino S, Lanteri-Minet M. Occipital nerve stimulation improves the quality of life in medically-intractable chronic cluster headache: Results of an observational prospective study. Cephalalgia. 2017 Oct;37(12):1173-1179. doi: 10.1177/0333102416673206. Epub 2016 Oct 3. PMID 27697849